CLINICAL TRIAL: NCT06907160
Title: A Prospective Cohort Study to Explore Biomarkers for Response to Neoadjuvant Chemoimmunotherapy in Stage II-III Non-small Cell Lung Cancer
Brief Title: Exploratory Biomarker Analysis of Neoadjuvant Chemoimmunotherapy Followed by Pulmonary Resection in Stage II-III Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-0434
Record Dates: First submitted 2024-12-04; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Clinical Stage II to III Non-Small Cell Lung Cancer
Keywords: NSCLC; Neoadjuvant chemoimmunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ·Before Neoadjuvant ICI treatment; 1) whole blood 20ml 2) Paraffin specimen from needle biopsy or bronchoscopy biopsy performed at the time of initial diagnosis and staging ·After Neoadjuvant ICI treatment 1) whole blood 20ml 2) One piece of tumor tissue sample (fresh tissue, 1cm x 1cm) scheduled to be discarded after surgery is collected on the day of surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant Immunotherapy: Establishment of a neoadjuvant ICI treatment cohort for resectable stage II-III lung cancer patients and acquisition of clinical-pathological-radiological data

SUMMARY:
1. To explore tissue-based biomarkers to select patients who do not respond to neoadjuvant immunotherapy (non-responders) at the point of diagnosis
2. To explore blood-based non-invasive biomarkers to predict pathological complete response (pCR) before surgery

DETAILED DESCRIPTION:
1. Construction of a neoadjuvant chemoimmuntherapy cohort of resectable stage 2-3 lung cancer patients and acquisition of clinical-pathological-radiological data.
2. Plasma from individual patient will be collected at preneoadjuvant and postneoadjuvant stages and ctDNA analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven clinical stage II-III lung cancer patients
* No driver mutations (EGFR mutation and ALK alteration)
* Whole body performance (ECOG) 0-1
* Those over 19 years of age
* Subject who submitted Informed consent form

Exclusion Criteria:

* Under 19 years of age
* If there is a history of causing infection or other serious medical problems that impair the patient's function and make it difficult to comply with the study protocol.
* Patients for whom the investigator determines that the patient should not participate in the clinical trial because the patient is judged to be unable to comply with the clinical trial procedures and requirements (a person lacking medical capacity)
* Other patients (pregnant women, etc.) determined by the clinical trial director to be unsuitable for this clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who visited the Severance Hospital Lung Cancer Center Outpatient Clinic (Thoracic Surgery and Hematology Oncology) where the research team is affiliated will be registered after reviewing whether they meet the above selection/exclusion criteria by a researcher assigned by the research director.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic response after surgery, assessed according to IASLC pathologic response criteria, including major pathologic response and pathologic complete response in resected specimens following neoadjuvant CIT. | Within the first 30 days (plus or minus 3 days) after surgery
  Pathologic response after surgery will be assessed according to the IASLC pathologic response criteria in resected tumor specimens following neoadjuvant CIT.
  Pathologic Complete Response (pCR): No residual viable tumor cells (0% viable tumor).
  Major Pathologic Response (MPR): ≤10% residual viable tumor cells. Evaluation Method: Pathologic response will be determined by histopathological examination of the resected tumor tissue, with tumor regression grading based on hematoxylin and eosin (H&E) staining.

SECONDARY OUTCOMES:
Progression-free survival | Defined as time from initiation of neoadjuvant therapy to first disease recurrence or death (whichever occurred first), assessed up to 36 months
  Defined as time from initiation of neoadjuvant therapy to first disease recurrence or death (whichever occurred first), assessed up to 36 months.
  Recurrence was defined as a diagnosis of metastatic disease, new locoregional disease, or any additional treatments for NSCLC after a 90-day treatment-free interval (to indicate the end of primary treatment and serve as a proxy for disease-free state postsurgery) starting right after initial surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided